CLINICAL TRIAL: NCT03561129
Title: Does the Operator Performing the Embryo Transfer Significantly Influence the Cycle Outcome: A Retrospective Evaluation of Humanitas Fertility Center's Experience
Brief Title: Embryotransfer Operator and Pregnancy Rate
Acronym: Operator
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: XXX/2018
Record Dates: First submitted 2018-06-07; First posted 2018-06-19 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Sterility
MeSH Terms: conditions — Infertility | interventions — Embryo Transfer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Embryo transfer — all the fresh embryo transfers, performed between January 1997 and December 2016 at Humanitas Fertility Center after IVF-ICSI cycles, divided per operator

SUMMARY:
Several studies had analyzed the correlation between embryo transfer operator experience and implantation, clinical pregnancy, abortion and delivery rate.

The aim of the present study is determining if the probabilities of embryo implantation and pregnancy are associated to the operator performing the embryo transfer.

This study allows following more than 30 different operators in a global period of 20 years with almost 20,000 procedures.

DETAILED DESCRIPTION:
Several studies had analyzed the correlation between embryo transfer operator experience and implantation, clinical pregnancy, abortion and delivery rate. Until now, the evidences are mixed and inconclusive.

The aim of the present study is determining if the probabilities of embryo implantation and pregnancy are associated to the operator performing the embryo transfer.

The database includes all the fresh embryo transfers, performed between January 1997 and December 2016 at Humanitas Fertility Center after IVF-ICSI cycles. Only embryo transfers performed by the surgeon on duty for that day ("Gynecologist of the Day") will be included.

Secondary end point is to evaluate if it is possible to draw a learning curve for transfer in terms of pregnancies for the different surgeons.

The strength of this study relies on the completeness of the preoperative factors and follow up and on the vastest dataset in literature that can permit to correct for multiple confounders and analyze a wide group of outcomes.

ELIGIBILITY:
Inclusion Criteria:

* fresh embryos' transfers
* embryo transfers performed only by the surgeon on duty for that day ("Gynecologist of the Day")

Exclusion Criteria:

* cryo thawed embryos' transfers

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study database includes all the fresh embryo transfers, performed between January 1997 and December 2016 at Humanitas Fertility Center after IVF-ICSI cycles. Only embryo transfers performed by the surgeon on duty for that day ("Gynecologist of the Day") will be included. A wider similar database was used for a previous research.
  Data are collected using an exclusive internal web-based database.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Actual)
Dates: Start 1997-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate per operator | 20 years
  number of viable intrauterine embryos/ total number of embryos transferred per operator

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uyar A, Bener A, Ciray HN, Bahceci M. Physician experience in performing embryo transfers may affect outcome. Fertil Steril. 2011 Apr;95(5):1860-2. doi: 10.1016/j.fertnstert.2010.10.036. PMID 21075368
- [Background] van Weering HG, Schats R, McDonnell J, Vink JM, Vermeiden JP, Hompes PG. The impact of the embryo transfer catheter on the pregnancy rate in IVF. Hum Reprod. 2002 Mar;17(3):666-70. doi: 10.1093/humrep/17.3.666. PMID 11870120
- [Derived] Cirillo F, Patrizio P, Baccini M, Morenghi E, Ronchetti C, Cafaro L, Zannoni E, Baggiani A, Levi-Setti PE. The human factor: does the operator performing the embryo transfer significantly impact the cycle outcome? Hum Reprod. 2020 Feb 29;35(2):275-282. doi: 10.1093/humrep/dez290. PMID 32100020